CLINICAL TRIAL: NCT03293446
Title: AC/DC Study: Acidification Test in Patients With Chronic Kidney Disease and Healthy Controls
Acronym: AC/DC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Ewout Hoorn, doctor, Erasmus Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NL57148.078.16
Record Dates: First submitted 2017-09-20; First posted 2017-09-26 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Chronic Kidney Disease stage4

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with chronic kidney disease (Experimental)
  Interventions: Diagnostic Test: Urinary acidification test
- Healthy controls (Active Comparator)
  Interventions: Diagnostic Test: Urinary acidification test

INTERVENTIONS:
Diagnostic Test: Urinary acidification test — Urinary acidification by administration of ammonium chloride (100 mg/kg body weight, given orally) during a single-day hospital admission.

SUMMARY:
In this study the effect of an acute acid load on the intrarenal renin angiotensin-system is evaluated in patients with chronic kidney disease and healthy controls

DETAILED DESCRIPTION:
Metabolic acidosis is one of the metabolic complications of chronic kidney disease (CKD). Correction of metabolic acidosis in CKD has been shown to prevent further loss of kidney function over time. Currently, a clinical trial (the BIC-study, MEC-2013-332) is conducted in which patients with CKD and metabolic acidosis receive sodium bicarbonate, sodium chloride, or no treatment (time control) to address the hypothesis that the beneficial effects of acidosis correction are mediated through inhibition of the intrarenal renin-angiotensin system (RAS). It is unknown, however, if and how acute changes in acid-base status affect the intrarenal RAS during CKD. In the present study it is hypothesized that an acute acid load increases the activity of the intrarenal RAS, and that this response is exaggerated in patients with CKD compared with healthy controls.

ELIGIBILITY:
Patients with CKD:

* Male or female adults (≥18 years)
* Chronic kidney disease stage 4 (eGFR: 15-30 ml/min/1.73 m2, calculated using the CKD-EPI equation)

Healthy controls:

* Healthy male or female adults (≥ 18 years)
* Normal kidney function (eGFR > 90 ml/min/1.73 m2, calculated using the CKD-EPI equation)

Exclusion Criteria:

* CKD patients
* Plasma bicarbonate level < 20.0 mmol/l
* Serum potassium >5.5 mmol/l
* Sodium bicarbonate use in the month preceding the test
* Heart failure (NYHA III or IV)
* Liver cirrhosis (Child Pugh B or C)
* Blood pressure >140/90 mmHg despite the use of 3 different anti-hypertensive drugs
* Kidney transplantation
* Use of calcineurin inhibitors (these immunosuppressive drugs affect acid-base balance)
* Known urea cycle disorder
* Alcoholism or drug use
* Pregnancy
* Current use of antibiotics, NSAIDS or alkalizing drugs (sodium-bicarbonate, citric acid, potassium citrate, acetazolamide)
* Inability to adhere to the study protocol (due to language barrier or intellectual disability)

Healthy controls:

* eGFR < 90 ml/min/1.73 m2 (calculated using the CKD-EPI equation)
* Plasma bicarbonate < 20 mmol/l
* History of, or drugs for, diabetes mellitus
* History of chronic diarrheal disease
* Ileostomy/colostomy
* Known urea cycle disorder
* Alcoholism or drug use
* Pregnancy
* Current use of antibiotics, antihypertensive drugs, NSAIDS or alkalizing drugs (sodium-bicarbonate, citric acid, potassium citrate, acetazolamide)
* Inability to adhere to the study protocol (due to language barrier or intellectual disability)

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — only males
Enrollment: 29 (Actual)
Dates: Start 2016-10-07 (Actual); Primary Completion 2018-11-11 (Actual); Study Completion 2018-11-11 (Actual)

PRIMARY OUTCOMES:
Urinary renin | up to 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided